CLINICAL TRIAL: NCT06011044
Title: Intercostal Nerve Block With Local Anesthesia Administered Via Incision-specific Multi-site Injection for Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bixin Wen (Other)
Responsible Party: Sponsor-Investigator, Bixin Wen, Principal Investigator, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bwen
Record Dates: First submitted 2023-06-22; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Intercostal Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal nerve block with ropivacaine（0.5%） (Experimental): This group of patients will be further divided into 2 groups. Group A (incision-specific multi-site injection) received intraoperative 3-8 intercostal nerve block with 0.5% ropivacaine. Group B (single injection) received intraoperative 3-5 intercostal nerve block with 0.5% .After completing lung surgery, fully exposing the lateral and posterior chest wall. From the inside view of the chest cavity, the intercostal nerve enters the correlated intercostal space between the posterior intercostal membrane and the parietal pleura. The needle of the 1ml syringe was held with a thoracoscopic ovale forceps and the target intercostal nerves were confirmed. It is only necessary to puncture the parietal pleura at the side of the intercostal nerve to perform the block. Inject ropivacaine(1ml, 0.5%) into the target nerve. At the same time, we recorded patients' mental status and vital signs to avoid systemic toxicity.
  Interventions: Procedure: Intercostal Nerve Block
- no intercostal nerve block. (No Intervention): This group of patients will not receive intraoperative intercostal nerve block with 0.5% ropivacaine. After completing lung surgery, fully exposing the lateral and posterior chest wall. From the inside view of the chest cavity, the intercostal nerve enters the correlated intercostal space between the posterior intercostal membrane and the parietal pleura. The needle of the 1ml syringe was held with a thoracoscopic ovale forceps and the target intercostal nerves were confirmed. Inject physiologic saline(1ml) into the target nerve.

INTERVENTIONS:
Procedure: Intercostal Nerve Block — The intercostal nerve block test is a medical intervention that involves the administration of a local anesthetic to the intercostal nerves, which are located between the ribs. The intervention involves injecting a small amount of anesthetic solution near the targeted intercostal nerves, which temporarily numbs the area and provides potential pain relief. The intercostal nerve block test is considered a diagnostic tool to help guide further treatment decisions for conditions such as intercostal neuralgia, rib fractures, or postoperative pain. It is generally a safe and well-tolerated procedure, often performed under local anesthesia or with the assistance of image guidance to ensure accurate needle placement. Following the test, the patient's response is evaluated, and if pain relief is achieved, it may indicate that intercostal nerve block injections could be an appropriate treatment option.
  Arms: Intercostal nerve block with ropivacaine（0.5%）

SUMMARY:
The goal of this clinical trial is to test analgesic effect of intercostal nerve block in different range. The main question it aims to answer are:

question 1: whther incision-specific multi-site injection (ISMSI, from the 3rd to 8th intercostal nerve) can improve the analgesic benefits .

The participants will be divided into three groups to compare the analgesic effects of different intercostal nerve blocks

DETAILED DESCRIPTION:
Postoperative pain after thoracic surgery is usually severe, and potentially leads to worse outcomes. It is well known that the use of intercostal nerve block (ICNB) analgesia with local anesthesia is common in thoracic surgery. Compared with the traditional standard of epidural analgesia, it has the advantages of less effect on respiratory or circulation system and less postoperative complications such as hypotension and hematoma. However, the details of ICNB form different hospital are in different ways. And it is unclear how many intercostal nerves should be blocked. And it is unknown which area should be payed more attention either, like the incision area or the chest tube port. It is hypothesized that the incision-specific multi-site injection (ISMSI, from the 3rd to 8th intercostal nerve) can improve the analgesic benefits due to cover area of both incision and chest tube port. To test this hypothesis, the investigators did this study to evaluate the analgesic effect of different ICNB methods.

The participants will be divided into three groups. A(incision-specific multi-site injection, received intraoperative 3-8 intercostal nerve block ) B(single injection, received intraoperative 3-5 intercostal nerve block ) and C(received no intercostal nerve block). Then compare the analgesic effects of the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery for small pulmonary nodules in the Department of Thoracic Surgery, China-Japan Friendship Hospital in Beijing
2. Age≥ 18 years old
3. Lung small nodules with a diameter of ≤ 2cm, pure ground-glass/mixed/solid nodules
4. Permanent residents can be followed up for a long time
5. Sign informed consent.

Exclusion Criteria:

1. Refusal to sign informed consent
2. Damaged heart, lung, liver and kidney function
3. Contraindications to surgery, such as inability to tolerate anesthesia, distant metastasis, bleeding tendency, etc c(4) Combined with severe emphysema, tuberculosis, pneumothorax, pleural effusion (5) Patients have other conditions that are not suitable for interventional surgery, such as pregnancy, lactation, long-term use of immunosuppressants, and serious infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-19 (Estimated); Primary Completion 2023-10-19 (Estimated); Study Completion 2023-10-19 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | first month after surgery
  We will use VAS score to assess the analgesic effects . The Visual Analogue Scale (VAS) has been in use for the measurement of intangible quantities such as pain since the 1920s. It consists of a line usually 100mm in length, with anchor descriptors such as "no pain" and "worst pain imaginable", The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm.

SECONDARY OUTCOMES:
The Visual Analogue Scale (VAS) | third month after surgery
  We will use VAS score to assess the analgesic effects . The Visual Analogue Scale (VAS) has been in use for the measurement of intangible quantities such as pain since the 1920s. It consists of a line usually 100mm in length, with anchor descriptors such as "no pain" and "worst pain imaginable", The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm.

IPD SHARING:
Plan to Share IPD: Undecided